CLINICAL TRIAL: NCT01651078
Title: Laser Ablation After Stereotactic Radiosurgery
Acronym: LAASR
Status: Completed | Type: Observational
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: LAASR
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Brain Tumors; Progression; Radiation Necrosis; Quality of Life
Keywords: Metastatic Brain Tumors; Progression; Radiation Necrosis; Quality of Life
MeSH Terms: conditions — Brain Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Main cohort: Patients with radiographic evidence of lesion regrowth following prior treatment with stereotactic radiosurgery (regardless of the process being suspected recurrent or progressive brain metastasis versus radiation necrosis) and who already scheduled for NeuroBlate procedure.

SUMMARY:
The need for new technologies and devices in the field of neurosurgery is well established. In April 2013, FDA cleared NeuroBlate™ System, minimally invasive robotic laser thermotherapy tool. It employs a pulsed surgical laser to deliver targeted energy to abnormal brain tissue caused by tumors and lesions. This post-marketing, multi-center study will include patients with metastatic tumors who failed stereotactic radiosurgery and are already scheduled for NeuroBlate procedure. The study will collect clinical outcome, Quality of Life (QoL) and, where feasible, healthcare utilization data for publication.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient has signed and received a copy of the Informed Consent Form
2. Patient may have up to 3 target supratentorial metastatic lesions previously treated with stereotactic radiosurgery, with radiological evidence of progression, pseudoprogression or radionecrosis. Subject may have additional non target lesions present as long as they are not expected (in Investigator's judgment) to contribute to symptomatology during the course of the study or confound interpretation of radiological and clinical measures.
3. Karnofsky Performance Status (KPS) ≥ 60.

Key Exclusion Criteria:

1. Females who are pregnant, breast feeding, or plan to become pregnant in the 6 months following index procedure.
2. Leptomeningeal metastases.
3. Uncontrolled infectious process.
4. Uncontrolled hypertension (systolic >180 mm Hg), angina pectoris, or cardiac dysrhythmia, or recent (within 6 weeks) history of intracranial hemorrhage.
5. Serious infection, immunosuppression or concurrent medical condition (chronic or acute in nature) that may prevent safe participation or ability to meet follow-up requirements.
6. Abnormal absolute neutrophil count (ANC<1000/mm), platelets (<100,000/mm) or the administration of antiplatelet agents (aspirin, plavix etc) or anticoagulation within 7 days prior to treatment.
7. Inadequate bone marrow, liver and renal function (e.g., total bilirubin > 1.5 x ULN; AST, ALT > 2.5 x ULN; alkaline phosphatase > 2.5 x ULN; serum creatinine > 1.5 x ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiographic evidence of lesion regrowth following prior treatment with radiosurgery (regardless of the process being suspected recurrent or progressive brain metastasis versus radionecrosis).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Chiang, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - Yale School of Medicine, New Haven, Connecticut
  - Kansas University Medical Center, Kansas City, Kansas
  - Washington University in St Louis, St Louis, Missouri
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Ahluwalia M, Barnett GH, Deng D, Tatter SB, Laxton AW, Mohammadi AM, Leuthardt E, Chamoun R, Judy K, Asher A, Essig M, Dietrich J, Chiang VL. Laser ablation after stereotactic radiosurgery: a multicenter prospective study in patients with metastatic brain tumors and radiation necrosis. J Neurosurg. 2019 Mar 1;130(3):804-811. doi: 10.3171/2017.11.JNS171273. Epub 2018 May 4. PMID 29726782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four (44) patients were enrolled between October 2012 and December 2015 across six centers in the United States (per the protocol, LAASR enrolled all patients who were scheduled to undergo a NeuroBlate procedure). Forty-two (42) patients underwent the procedure and were followed under the protocol as the "NeuroBlate Procedure" treatment arm.
Groups:
- NeuroBlate Procedure: Patients with radiographic evidence of lesion regrowth following prior treatment with stereotactic radiosurgery (regardless of the process being suspected recurrent or progressive brain metastasis versus radiation necrosis) and who underwent the NeuroBlate procedure
Period: Overall Study
Arm/Group | NeuroBlate Procedure
Started | 42 (Two (2) out of 44 patients were enrolled but did not go on to have the NeuroBlate Procedure.)
Completed | 16
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Main Cohort
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 60 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 42
Biopsy-confirmed radiation necrosis or metastatic brain tumor [Number; unit: patients] | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Progression-Free Survival (PFS)
Description: To describe local (CNS) progression-free survival rate in patients with failed radiosurgery for brain metastases treated with the NeuroBlate System. Sites were requested to submit imaging to a centralized core laboratory for analysis. A total of 27 patients had images submitted--27/42 (64%) of patients submitted follow-up images at 12-weeks and 16/42 (38%) patients submitted follow-up imaging at 26 weeks. Due to the low submission of follow-up images at 26-weeks, 12-weeks and last follow-up are reported.
Time Frame: Images were collected at 12 and 26 weeks post index procedure.
Population: Sites were requested to submit imaging to a centralized core laboratory for analysis. A total of 27 patients had images submitted--27/42 (64%) of patients submitted follow-up images at 12-weeks and 16/42 (38%) patients submitted follow-up imaging at 26 weeks.
Measure: Number; unit: percentage of patients
Groups:
- NeuroBlate Procedure: Patients with radiographic evidence of lesion regrowth following prior treatment with stereotactic radiosurgery (regardless of the process being suspected recurrent or progressive brain metastasis versus radiation necrosis) and who already scheduled for NeuroBlate procedure.
Arm/Group | NeuroBlate Procedure
Number analyzed (Participants) | 27
percentage of patients
  12-weeks | 74
  Last Follow-up | 74

2. Secondary Outcome: Quality of Life (Change in The Functional Assessment of Cancer Therapy-Brain (FACT-Br) Score.
Description: FACT-Br questionnaire sub-scores (Physical well-being, social/family well-being, emotional well-being, functional well-being, brain cancer subscale) are summed together, leading to a FACT-Br total score on a scale from 0-200; larger scores indicate better overall quality of life. This outcome measured the FACT-Br score change from Baseline at both 12 and 26 weeks post NeuroBlate procedure (values at 12 and 26 weeks, respectively, minus value at baseline). Version 4 of the Fact-BR scoring guidelines were used.
Time Frame: baseline, 12 and 26 weeks post index procedure
Population: Due to study attrition, the full cohort was unavailable for analysis.
Measure: Median (Full Range); unit: change in FACT-Br score
Arm/Group | NeuroBlate Procedure
Number analyzed (Participants) | 42
change in FACT-Br score
  Change in 12-week FACT-Br from Baseline: number analyzed (Participants) | 27
  Change in 12-week FACT-Br from Baseline | 3.8 [-71.8 to 40]
  Change in 26-week FACT-Br from Baseline: number analyzed (Participants) | 16
  Change in 26-week FACT-Br from Baseline | 7.0 [-34.7 to 34.3]

3. Secondary Outcome: Overall Survival
Description: To describe/estimate the overall survival after the NeuroBlate Procedure.
Time Frame: 12 and 26 weeks post index procedure
Measure: Number; unit: percentage of patients
Arm/Group | NeuroBlate Procedure
Number analyzed (Participants) | 42
percentage of patients
  12-week Kaplan-Meier survival | 86.5
  26-week Kaplan-Meier survival | 72.2

4. Secondary Outcome: Percentage of Patients With Laser Ablation Related Adverse Events
Description: To continue to monitor factors impacting the safe and efficacious use of NeuroBlate
Time Frame: All adverse events reported through 26 weeks post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | NeuroBlate Procedure
Number analyzed (Participants) | 42
Participants
  Serious events associated with NeuroBlate | 0
  Non-serious events associated with NeuroBlate | 5
  No NeuroBlate-related adverse event | 37

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of patient consent (prior to the surgical procedure) to study withdraw/completion, up to 26 weeks.
Description: Events adjudicated as surgery- or LITT- associated are described in the adverse events section.
Arm/Group | Main Cohort
All-Cause Mortality (participants affected / at risk) | 8/42
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=42)
Pulmonary or other air embolism (Surgical and medical procedures) | 2 (2)
Seizures (Nervous system disorders) | 2 (2)
Hypotension (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations are discussed by the physicians in the full publication of the LAASR study data (open access): http://thejns.org/doi/pdf/10.3171/2017.11.JNS171273

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No